CLINICAL TRIAL: NCT06080165
Title: A Randomized Controlled Double-Blind Trial of Sirolimus for Improving Social Abilities in People With PTEN Germline Mutations
Brief Title: Sirolimus for Improving Social Abilities in People With PTEN Germline Mutations
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Investigator decided not to proceed with the trial.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-72157
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: PTEN Gene Mutation; PTEN Hamartoma Tumor Syndrome; PTEN Hamartoma Syndrome
Keywords: Sirolimus; Rapamune
MeSH Terms: conditions — Hamartoma Syndrome, Multiple | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus (Experimental): Participants that are 5 to 12.99 years old will start at 1 mg/m2/dose. Participants that are 13 to 45.99 years old and < 39.99 kg in weight will also start on 1 mg/day. Participants that are 13 to 45.99 years old and > 40 kg in weight will start on 2 mg/day. The target blood level will be 5-15 ng/ml with dose adjustment based on sirolimus levels obtained every 2 to 3 weeks after every dose change.
  Interventions: Drug: Sirolimus
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus — Experimental: Sirolimus Participants that are 5 to 12.99 years old will start at 1 mg/m2/dose. Participants that are 13 to 45.99 years old and < 39.99 kg in weight will also start on 1 mg/day. Participants that are 13 to 45.99 years old and > 40 kg in weight will start on 2 mg/day. The target blood level will be 5-15 ng/ml with dose adjustment based on clinical labs of sirolimus levels. The target blood level will be 5-15 ng/ml with dose adjustment based on sirolimus levels obtained every 2 to 3 weeks after every dose change.
  Other Names: Rapamune
  Arms: Sirolimus
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
The goal of this study is to examine the safety and treatment effects of sirolimus for targeting social communication deficits in people with genetic disorders associated with PTEN germline mutations, which are often referred to as PTEN Harmartoma Tumor Syndrome (PHTS). The mechanism of sirolimus in the body has shown promise for helping to improve social communication skills in case reports of people with PHTS. Everolimus, a closely related compound, also showed benefits in social communication skills in a previous pilot trial in people with PHTS. This is a 6 month double-blind trial followed by at 6 month open label extension trial.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: All participants will meet the following selection criteria:
* Male or female outpatients between 5.00 and 45.99 years of age
* PHTS confirmed by genetic testing;
* Fluent in English
* at least moderate severity of social skill deficits based on a social responsiveness scale t score ≥ 60
* Stable psychotropic and anti-epileptic medications for at least 4 weeks with the exception of fluoxetine which should be stable for at least 8 weeks
* Adequate Liver function (SGOT, SGPT, TBili, Alk Phos all<3x normal); HCT>27%; WBC > 3.0, ANC >1,500, and platelets >100,000
* adequate renal function with a GFR ≥ 50 ml/min/m2 as determined by the Schwartz Formula for children and MDRD for adults (www.nkdep.nih.gov/professionals/gfr_calculators/index)
* Negative urine pregnancy test for females and no plans to become pregnant or conceive a child while participating in the study. The effects of mTOR inhibitors on the developing fetus at the doses used in this study are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of the study. Because of the possibility of drug interactions and the potential effect of female hormones on the growth of kidney angiomyolipomas and lymphangioleiomyomatosis, estrogen-containing oral contraceptives are not recommended in women enrolled in this study, so an effective non-estrogen or barrier method of contraception must be used.
* Medically stable with no active medical problems such as unstable seizures or cardiovascular disease or cancer that is not in remission as evidenced by medical history; -No anticipated changes in frequency and intensity of existing interventions such as behavioral and developmental treatments, in home services, or speech therapy;
* No planned changes in school placement in children and adolescents;
* Availability of reliable transportation to attend clinic visits;
* availability of a trustworthy informant who interacts with subject on a regular basis;
* Ability to participate in the testing procedures to the extent that valid standard scores and biological samples can be obtained.

Exclusion Criteria:

* Participants will be excluded if one of the following is met:
* Significant medical illness, such as endocrinopathies, cardiovascular disease, or severe chronic malnutrition;
* Pregnancy, planned pregnancy, or unwillingness to use adequate contraception;
* Planned changes to concomitant medications;
* Concomitant therapy, or prior use within 3 months of the baseline visit, with an agent with known or possible anti-mTOR activity or concomitant therapy with strong inhibitors (e.g., cyclosporine and ketoconazole) or inducers of CYP3A;
* Active infection at time of enrollment;
* Participation in a clinical trial in the 30 days prior to study entry;
* Major surgery, radiation therapy or stereotactic radio-surgery within previous 4 weeks at time of enrollment; and
* Neurosurgery within prior 6 months at time of enrollment.

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in parent rated Social Responsiveness Scale, Second Edition Total Scores (SRS-2) total scores during treatment. | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6

SECONDARY OUTCOMES:
Clinical Global Impression Improvement (CGI-I) Scale changes during treatment. | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Change from baseline on parent rated Stanford Social Dimensions Scale (SSDS) | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6

OTHER OUTCOMES:
Change from baseline on Brief Observation of Social Communication Change (BOSCC) | Month 6
Change from baseline on Neurobehavioral Evaluation Tool (NET) Social Communication and Interaction subscale | Month 3, Month 6
Change from baseline on the Reading the Mind in the Eyes Test (RMET) | Month 6
Change from baseline on Purdue Pegboard (PP) Test | Month 6
Change from baseline on parent rated Dimensional Assessment of Restricted/Repetitive Behaviors (DARB) | Month 3, Month 6
Change from baseline on Vineland Adaptive Behavior Scales (VABS-III) | Month 3, Month 6
Change from baseline on Wide Range Assessment of Memory and Learning-2 (WRAML-2) | Month 6
Change from baseline on Clinical Global Impression Improvement (CGI-I) Scale changes during treatment. | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Change from baseline on parent reported Child or Adult Behavioral Checklist | Month 3, Month 6
Change from baseline on complete blood count (CBC) with differential as measured by peripheral blood | Month 1, Month 3, Month 5, Month 6
Change from baseline on comprehensive metabolic panel as measured by peripheral blood | Month 1, Month 3, Month 5, Month 6
Change from baseline on lipid profile as measured by peripheral blood. | Month 1, Month 3, Month 5, Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Data will be on the National Institute of Mental Health Data Archive (NDA).
Time Frame: shared twice per year
URL: https://nda.nih.gov/